CLINICAL TRIAL: NCT00993304
Title: A Trial to Assess the Effect of Liraglutide on Postprandial Triglyceride Levels in Subjects With Type 2 Diabetes
Brief Title: A Trial to Assess the Effect of Liraglutide on Blood Triglyceride (Fat) Levels After a Meal in Type 2 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-3534; 2008-003229-18 (EudraCT Number); U1111-1111-9161 (Other: WHO)
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: liraglutide
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — In the first 3-week period, the treatment will be one week with 0.6 mg, one week with 1.2 mg and one week with 1.8 mg liraglutide. Subsequently, a wash-out period of 3 to 9 weeks occurs and then a second period of 3 weeks' treatment with placebo. At the end of each of the 2 treatment periods, a high fat meal test will be performed.
  Arms: A
Drug: placebo — In the first 3-week period, the treatment will be with placebo. Subsequently, a wash-out period of 3 to 9 weeks occurs and then a second period of one week with 0.6 mg, one week with 1.2 mg and one week with 1.8 mg of liraglutide. At the end of each of the 2 treatment periods, a high fat meal test will be performed.
  Arms: B

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate whether a new compound, liraglutide, reduces the level of lipids (fat), including cholesterol, in the blood of type 2 diabetics, following a meal with high fat content.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus (diet and exercise treated, or treated with specific oral antidiabetics (metformin, sulfonylureas and glinides) mono- or combination therapy) diagnosed at least 3 months previously
* BMI between 18.5 and 40 kg/m2
* HbA1c between 6.5 and 10.0% both inclusive

Exclusion Criteria:

* Known or suspected allergy to trial products or related products
* Previous participation in this trial (randomised). Re-screening of screening failures is allowed only once
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptives are defined as combination oral contraceptives (OC), hormonal intra uterine devices (IUDs), implants and injectables; for Germany, a condom for the male partner must be used in combination with OC, IUD, implant or injectables for the duration of the trial and for 30 days following the last dose of trial medication) if not sterile or post-menopausal
* The receipt of any investigational drug within 3 months prior to this trial
* Previous insulin treatment (short-term insulin treatment of up to 7 days are exempted if this has occurred no later than 3 months prior to screening).
* Cancer (except basal cell skin cancer or squamous cell skin cancer) or any clinically significant disorder (except type 2 diabetes)
* Clinically significant active cardiovascular disease including history of myocardial infarction (heart attack) within the past 6 months and/or heart failure at the discretion of the Investigator.
* History of alcoholism or drug abuse during the last 12 months
* Blood donation within the last 3 months. Plasma donation within the last month.
* Additional exclusion criteria for Germany: Male subjects who are sexually active and have partners who are or could be pregnant, not using a barrier method of contraception (e.g. condom) for the duration of the trial and for 30 days following the last dose of trial medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
AUC0-8h (triglyceride), the area under the triglyceride-concentration-time curve in the interval 0-8 hours following a meal with a high fat content | after 3 weeks of treatment

SECONDARY OUTCOMES:
FFA (Free Fatty Acid), VLDL (Very Low Density), and apoB48: AUC0-8 hours after meal with a high fat content | after 3 weeks of treatment
Glucose, insulin, C-peptide and glucagon: AUC0-8 hours after meal with a high fat content | after 3 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Aarhus C, Denmark

REFERENCES:
- [Result] Hermansen K, Baekdal TA, During M, Pietraszek A, Mortensen LS, Jorgensen H, Flint A. Liraglutide suppresses postprandial triglyceride and apolipoprotein B48 elevations after a fat-rich meal in patients with type 2 diabetes: a randomized, double-blind, placebo-controlled, cross-over trial. Diabetes Obes Metab. 2013 Nov;15(11):1040-8. doi: 10.1111/dom.12133. Epub 2013 Jun 11. PMID 23683069
- [Result] Roge RM, Klim S, Ingwersen SH, Kjellsson MC, Kristensen NR. The Effects of a GLP-1 Analog on Glucose Homeostasis in Type 2 Diabetes Mellitus Quantified by an Integrated Glucose Insulin Model. CPT Pharmacometrics Syst Pharmacol. 2015 Jan;4(1):e00011. doi: 10.1002/psp4.11. Epub 2014 Dec 30. PMID 26225223
- [Derived] Petri KC, Jacobsen LV, Klein DJ. Comparable liraglutide pharmacokinetics in pediatric and adult populations with type 2 diabetes: a population pharmacokinetic analysis. Clin Pharmacokinet. 2015 Jun;54(6):663-70. doi: 10.1007/s40262-014-0229-z. PMID 25603819
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com